CLINICAL TRIAL: NCT01920633
Title: A Screening Protocol to Assess Adult and Adolescent Individuals With Down Syndrome for Eligibility to Participate in an Upcoming Study to Evaluate the Efficacy, Safety and Tolerability of RG1662 (Study BP27832)
Brief Title: A Screening Protocol to Assess Adults and Adolescents With Down Syndrome for Eligibility For Upcoming Study of RG1662 (Study BP27832)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BP28947; 2013-001264-33 (EudraCT Number)
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- People with Down syndrome

SUMMARY:
This is a single visit study in which people with Down syndrome aged 12-30 will attend the clinical center to undergo assessments to evaluate their eligibility for potential enrollment in the future BP27832 Phase II clinical study which will evaluate the efficacy, safety and tolerability of RG1662. Study participants may withdraw from this study at any time and for any reason.

ELIGIBILITY:
Inclusion Criteria:

Study participants will be assessed on the following criteria that they will be required to meet in order to participate in the future Phase II study BP27832:

* Males and females 12-30 years of age (18-30 in the US)
* Clinical diagnosis of Down syndrome (trisomy 21) documented by chromosomal analysis (karyotyping)
* Body-mass Index (BMI) 18-42 and 15-32 kg/m2 inclusive for adults and adolescents respectively
* Ability to complete the Clinical Evaluation of Language Fundamentals (CELF)-preschool 2 word classes task (i.e., ≥ 7 for the adults or ≥ 4 for the adolescents in the expressive raw score).
* Study participant willing and assenting or consenting to participate
* Parent or guardian willing to give written informed consent
* Study participants must have a parent, or other reliable caregiver who will agree to accompany the study participant to clinic visits during the treatment study, BP27832
* The parent or caregiver must be a constant and reliable informant with sufficient contact with the study participant to have detailed knowledge of the study participant's adaptive functioning in order to be able to complete assessments accurately
* Study participants must be verbal and able to be understood most of the time and must not use other forms of communication, signs, symbol boards or devices as their primary form of communication
* Study participants must have sufficient vision and hearing to participate in study evaluations
* Study participants on anti-epileptic treatment must be on stable doses for 4 weeks prior to enrollment in the treatment protocol

Exclusion Criteria:

In the future Phase II study, study participants must not meet any of the following criteria :

* Study participants with severe lactose intolerance
* Study participants with moderate or severe Obstructive Sleep Apnea (OSA) as defined by Apnea-Hypopnea Index (AHI) (>15 events per hour not well controlled by positive airway pressure therapy with stable settings) for 6 weeks prior to the screening visit
* Study participants with history of malignancy if not considered likely to be cured
* Personal history of infantile spasms, of epilepsy, of severe head trauma or Central Nervous System (CNS) infections (e.g. meningitis), with the exception of a single isolated febrile seizure
* Study participants with history of epilepsy within the last 2 years.
* Evidence of active, clinically significant, and unstable gastrointestinal, renal, hepatic, endocrine or cardiovascular system disease
* Study participants with a current Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosis of any primary psychiatric diagnosis (including autism spectrum disorder). Diagnoses that are secondary, such as intellectual disability, attention deficit hyperactivity disorder, depression and conduct disorder are allowed as long as they are considered stable and to not interfere with conduct of a future treatment study
* Study participants with a history of suicide attempt or deliberate self-harm due to suicidal ideation will not be included. Suicidal ideation (even in the absence of suicide attempt or deliberate self-harm) during the 6 months prior to screening
* Concomitant use of excluded approved or unapproved medications
* Personal or family history of congenital long QT syndrome
* History of hepatitis C or known Human Immunodeficiency Virus (HIV) infection
* Pregnant or breast feeding

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: People with Down syndrome
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2013-10-31 (Actual); Primary Completion 2015-01-31 (Actual); Study Completion 2015-01-31 (Actual)

PRIMARY OUTCOMES:
Identification of people with Down syndrome aged 12-30 eligible for upcoming BP27832 study of RG1662 | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (9):
  - Univ of CA San Diego; Neurosciences Comp.Alzheimer's, La Jolla, California
  - Emory University School of Medicine; Department of Human Genetics & Pediatrics, Decatur, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital., Baltimore, Maryland
  - Massachusette General Hospital; Medical Genetics, Boston, Massachusetts
  - Duke Clin Rsch Institute, Durham, North Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Utah School of Medicine; Department of Pediatrics, Salt Lake City, Utah
  - University of Wisconsin Madison, Waisman Center, Madison, Wisconsin
- Argentina (2):
  - Instituto de Investigaciones Neurologicas Raul Carrea FLENI, Capital Federal
  - Instituto Neurologia Bs As, Ciudad Autonoma de Bs As
- True North Clinical Research Kentville, Kentville, Nova Scotia, Canada
- Mexico (3):
  - Hospital Dr. Angel Leaño; Pediatria, Guadalajara, Jalisco
  - Clínica Para la Atención del Neurodesarrollo, Aguascalientes
  - Hospital Médica Tec 100, Querétaro
- New Zealand (3):
  - Auckland Clinical Studies, Auckland
  - University of Otago; Psychological Medicine Department, Dunedin
  - Wellington Hospital Research Office, Wellington
- KK Women's and Children's Hospital; Department of Neonatology, Singapore, Singapore
- Spain (3):
  - UVaMID Hospital Santa Caterina;; Servicio de Neurología, Salt, Girona
  - IMIM, Human Pharmacology and Clinical Neurosciences,, Barcelona
  - Hospital Universitario de la Princesa; Medicina Interna, Madrid